CLINICAL TRIAL: NCT00702910
Title: A Randomised, Single-dose, Double-blind, Placebo-controlled, 5-way Crossover Study to Investigate the Efficacy, Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Inhaled Doses of GW642444M With and Without Magnesium Stearate in Asthmatic Patients
Brief Title: A Study to Investigate the Effect of Inhaling Single Doses of Different Formulations of GW642444M in Asthmatic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: B2C111401
Record Dates: First submitted 2008-06-18; First posted 2008-06-20 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Asthma patients; Magnesium stearate; Tolerability; Safety; Lactose; GW642444M; Pharmacodynamics; Efficacy; Pharmacokinetics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — stearic acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- GW642444M/lactose (Experimental): GW642444M/lactose 6.25, 25 and 100 microgram, single inhaled dose for two days treatment in each treatment sequence (crossover design)
  Interventions: Drug: Placebo; Drug: GW642444; Drug: Magnesium Stearate
- GW642444M/MgSt (Experimental): GW642444M/MgSt 6.25, 25 and 100 microgram, single inhaled dose for two days treatment in each treatment sequence (crossover design)
  Interventions: Drug: Placebo; Drug: GW642444; Drug: Magnesium Stearate
- Placebo (Placebo Comparator): Placebo containing lactose, single inhaled dose for two days treatment in each treatment sequence (crossover design)
  Interventions: Drug: Placebo; Drug: GW642444; Drug: Magnesium Stearate

INTERVENTIONS:
Drug: Placebo — comparator
Drug: GW642444 — investigational drug or placebo
  Other Names: Placebo
Drug: Magnesium Stearate — Magnesium Stearate

SUMMARY:
This study will involve the use of a new medicine called GW642444 being developed for the treatment of asthma and chronic obstructive pulmonary disease (COPD). The purpose of the study is to see how safe and how well tolerated the study drug is when inhaled in two different formulations as a fine powder by asthmatic patients. In addition, the study is designed to examine the effect of the study drug on the lungs, how the study drug affects parts of the body other than the lungs and to see how the body affects the study drug when it is given in single doses.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a documented history of persistent asthma, with the exclusion of other significant pulmonary diseases (e.g. chronic bronchitis, emphysema, bronchiectasis, cystic fibrosis or bronchopulmonary dysplasia).
* Male subjects or female subjects aged between 18 to 70 years.
* A female subject is eligible to participate if she is of:

  * Non-childbearing potential defined as pre-menopausal females with a documented tubal ligation or hysterectomy; or postmenopausal defined as 12 months of spontaneous amenorrhea [in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) > 40 MlU/ml and estradiol < 40 pg/ml (< 140 pmol/L) is confirmatory.
  * Child-bearing potential and agrees to use one of the contraception methods listed in Section 8.1 for an appropriate period of time (as determined by the product label or investigator) prior to the start of dosing to sufficiently minimize the risk of pregnancy at that point. Female subjects must agree to use contraception until 2 days post last-dose.
* Subjects who are current non-smokers, who have not used any inhaled tobacco products (snuff is permitted) in the 12 month period preceding the screening visit and who have a pack history of ≤ 10 pack years.
* Subjects with clinically stable, mild to moderate persistent asthma within the 4 weeks preceding the screening visit and with a screening pre-bronchodilator FEV1 ≥ 60 % predicted as defined in the GINA guidelines [Global Initiative for Asthma (GINA), 2006] (having abstained from bronchodilators for the required period). Predicted values are based on the ECCS 1993 normal ranges.
* Body weight ≥ 50 kg and body mass index (BMI) within the range 19 - 29.9 kg/m2
* During the screening visit, subjects must demonstrate the presence of reversible airway disease, defined as an increase in FEV1 of ≥ 12.0% over baseline and an absolute change of ≥ 200 mL within 30 minutes following a single 400 mcg salbutamol dose.
* ECG criteria as per protocol
* Subjects who are currently taking ICS at a total daily dose of 200 to 500 mcg of FP or equivalent ICS.
* Subjects who are able and willing to give written informed consent to take part in the study.

Exclusion Criteria:

* Subjects who have a past or present disease, which as judged by the Investigator and the Medical Monitor, which may affect the safety of the subject or outcome of this study.
* A screening Holter ECG tracing that reveals clinically concerning arrhythmias.
* Subjects who have suffered an upper or lower respiratory tract infection within 4 weeks of the screening visit
* Subjects with a history of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with either respiratory arrest or hypoxic seizures.
* Asthma exacerbations requiring treatment with oral corticosteroids: any exacerbations within 3 months of the screening visit or two or more exacerbations within 6 months of the screening visit or admittance to hospital for an asthma exacerbation within 1 year of the screening visit.
* Subjects classified as suffering from severe asthma as defined by the ATS guidelines
* Subjects who have taken high doses of an inhaled corticosteroid (> 500 mcg FP/day or equivalent) within 8 weeks of the screening visit or oral steroids within 12 weeks of the screening visit.
* Subjects who have changed their inhaled corticosteroid treatment within the last 6 weeks before screening or can be expected to do so during the study.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four NCE's within 12 months prior to the first dosing day
* Any adverse reaction including immediate or delayed hypersensitivity to any β2 agonist or sympathomimetic drug, or known or suspected sensitivity to the constituents of GW642444 inhalation powder (e.g., lactose, milk protein, magnesium stearate).
* Subjects with a positive pre-study Hepatitis B surface antigen, positive Hepatitis C antibody or HIV result (if tested as per site SOPs) within 3 months of the start of the study.
* Neurological or psychiatric disease or history of drug or alcohol abuse which would interfere with the subject's proper completion of the protocol requirements, including compliance.
* Abuse of alcohol is defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units (males) or defined as an average weekly intake of greater than 14 units or an average daily intake of greater than 2 units (females).
* 1 unit is equivalent to a half pint (220 mL) of beer or 1 measure (25 mL) of spirits or 1 glass (125 mL) of wine.
* The subject has a positive pre-study urine drug test screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* The subject has a positive pre-study alcohol or smoking breath or urinary test.
* Where participation in the study would result in donation of blood in excess of 500 mL within a 56 day period.
* Subjects with clinically relevant findings on laboratory safety tests.
* Subjects with laboratory values outside the reference range may be included if the Investigator and medical monitor agree that these findings would not put the subject at risk or interfere with the objectives of the study.
* Subjects with known hypersensitivity to salbutamol or any ingredient in this preparation
* Subjects who have taken P-gp inhibitors and CYP 450 3A4 inhibitors (e.g. Ketoconazole) within 6 weeks or theophyllines within 2 weeks of the screening visit.
* Inability to use the novel dry powder inhaler.
* Pregnant females as determined by positive hCG (serum or urine) test at screening or prior to dosing.
* Lactating females.
* Unwillingness or inability to follow the procedures outlined in the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-04-27 (Actual); Primary Completion 2008-10-04 (Actual); Study Completion 2008-10-04 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline (pre-dose) FEV1 in trough (mean of the FEV1 values obtained 23 and 24 hours after dosing) FEV1 | on going

SECONDARY OUTCOMES:
Mean change from baseline (pre-dose) in FEV1 (i.e. derive separate responses for each FEV1 obtained over 24 hours after dosing). | on going
General safety and tolerability, including adverse events, laboratory safety tests (haematology, clinical chemistry and urinalysis), vital signs and, 12-lead ECG. | on going
Weighted mean and maximum value (0 - 4 h) QTc(B) | on going
Weighted mean and maximum value (0 - 4 h) QTc(F) | on going
Weighted mean and maximum value (0 - 4 h) supine heart rate | on going
Weighted mean and maximum value (0 - 4 h) supine systolic blood pressure | on going
Weighted mean and minimum value (0 - 4 h) supine diastolic blood pressure | on going
Weighted mean and maximum value glucose (0 - 4 h) | on going
Weighted mean and minimum value potassium (0 - 4 h) | on going
Single dose derived plasma pharmacokinetic parameters (AUC(0-t), Cmax, tmax) for GW642444 and GI179710 (triphenylacetate counterion) | on going
Estimate GW642444 concentration (Cmax) -systemic pharmacodynamic relationship for PD parameters, including heart rate, potassium & glucose levels | on going

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- Australia (2):
  - GSK Investigational Site, Auchenflower, Queensland
  - GSK Investigational Site, Clayton, Victoria
- GSK Investigational Site, Wellington, New Zealand

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Kempsford R, Norris V, Siederer S. Vilanterol trifenatate, a novel inhaled long-acting beta2 adrenoceptor agonist, is well tolerated in healthy subjects and demonstrates prolonged bronchodilation in subjects with asthma and COPD. Pulm Pharmacol Ther. 2013 Apr;26(2):256-64. doi: 10.1016/j.pupt.2012.12.001. Epub 2012 Dec 8. PMID 23232038
- See also: Results for study B2C111401 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/B2C111401?search=study&search_terms=B2C111401#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: B2C111401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2C111401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: B2C111401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2C111401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2C111401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C111401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2C111401 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register